CLINICAL TRIAL: NCT01561859
Title: Brain Imaging, Cognitive Enhancement and Early Schizophrenia
Acronym: BICEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Pittsburgh (Other); Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matcheri S. Keshavan MD, Stanley Cobb Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011P000267; R01MH092440 (NIH)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Early Course Schizophrenia; Cognitive Enhancement Therapy; Enriched Supportive Therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive enhancement therapy (Experimental): Cognitive Enhancement Therapy (CET) consists of approximately 60 hours of computer-assisted neurocognitive training in attention, memory, and problem-solving; and 45 social-cognitive group sessions that employ in vivo learning experiences to foster the development of social wisdom and success in interpersonal interactions. CET begins with 3 months of weekly 1-hour neurocognitive training in attention, after which patients begin the weekly 1.5-hour social-cognitive groups. Neurocognitive training then proceeds concurrently with the socialcognitive groups
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Enriched Supportive Therapy (Active Comparator): Enriched Supportive Therapy is an individual approach that includes the established principles of supportive therapy previously tested by our group, which are "enriched" by selected practice principles from the effective Personal Therapy. These manualized supportive therapeutic practices include active listening, correct empathy, appropriate reassurance, basic psychoeducation, including computer-based educational programs, reinforcement of health-promoting initiatives, the provision of case management, and reliance on the advocacy and advice of the therapist in times of crisis.
  Interventions: Behavioral: Enriched Supportive Therapy

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — Cognitive Enhancement Therapy (CET) consists of approximately 60 hours of computer-assisted neurocognitive training in attention, memory, and problem-solving; and 45 social-cognitive group sessions that employ in vivo learning experiences to foster the development of social wisdom and success in interpersonal interactions. CET begins with 3 months of weekly 1-hour neurocognitive training in attention, after which patients begin the weekly 1.5-hour social-cognitive groups. Neurocognitive training then proceeds concurrently with the socialcognitive groups.
  Arms: Cognitive enhancement therapy
Behavioral: Enriched Supportive Therapy — Enriched Supportive Therapy is an individual approach that includes the established principles of supportive therapy previously tested by our group, which are "enriched" by selected practice principles from the effective Personal Therapy. These manualized supportive therapeutic practices include active listening, correct empathy, appropriate reassurance, basic psychoeducation, including computer-based educational programs, reinforcement of health-promoting initiatives, the provision of case management, and reliance on the advocacy and advice of the therapist in times of crisis.
  Arms: Enriched Supportive Therapy

SUMMARY:
The proposed project is designed to examine the effects of cognitive rehabilitation on brain structure and function in a randomized trial of 102 early course schizophrenia patients treated for 18 months with either cognitive enhancement therapy (CET) or an Enriched Supportive Therapy (EST) control, and then followed-up at 1-year post-treatment.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and highly disabling disorder, making it imperative to apply interventions that alter its deleterious effects as early as possible. Impairments in neurocognition and social cognition, which appear to be linked to impaired structural and functional integrity in key brain regions, are the strongest predictors of functional disability in early course schizophrenia,making them key targets for early intervention. Although pharmacologic treatment of cognitive impairments is currently limited,our studies and others, including meta-analyses have shown that cognitive rehabilitation can be effective for addressing cognitive impairment in chronic patients. Most notably, Cognitive Enhancement Therapy (CET), a unique integrated approach to the rehabilitation of social and non-social cognitive impairments developed and tested by Hogarty and colleagues in our group, has shown substantial and lasting effects in chronic schizophrenia patients. Recently, the investigators have shown that the beneficial effects of CET can be successfully extended to those in the early phase of the disorder, resulting in large functional improvements.

The investigators have posited that CET can be particularly effective as an early intervention strategy by capitalizing on a fronto-temporal plasticity reserve, and the investigators are now observing compelling, albeit preliminary evidence that CET can indeed slow the progression of gray matter loss in these very regions of the brain, which is associated with significantly improved cognition (see Preliminary Studies). Preserved structural integrity and improved brain function in fronto-temporal regions may be the critical mechanisms for supporting cognitive improvement in early course schizophrenia, yet remarkably little is known about the neurobiologic effects of cognitive rehabilitation, the durability of these effects post-treatment, and whether an initial fronto-temporal reserve portends a greater treatment response. Our exciting preliminary findings of the neuroprotective effects of CET represent the first study to demonstrate that the structural integrity of the brain in the early course of schizophrenia can be altered using cognitive rehabilitation. It is critical that these morphologic findings are examined with more advanced imaging techniques in larger samples to gain a precise understanding of the underlying neurobiologic mechanisms and predictors of cognitive and functional enhancement in early course schizophrenia. These goals are reflective of the strategic plan of NIMH to identify underlying neural mechanisms of mental disorders that can facilitate treatment, and personalize care to optimize treatment response. To accomplish this, the investigators propose to use comprehensive structural and functional imaging methods to study 102 new early course schizophrenia patients treated for 18 months in a randomized trial of CET or Enriched Supportive Therapy (EST) and: Aim #1: Confirm the neuroprotective effects of CET on fronto-temporal brain structure. Structural magnetic resonance imaging (MRI) assessments will be collected along with cognitive and functional outcome data at baseline, 9, and 18 months. It is hypothesized that patients treated with CET will demonstrate decreased loss of fronto-temporal gray matter relative to EST, and that this neuroprotection will be a mechanism of cognitive and functional improvement. Effects on other key brain regions will also be explored; Aim #2: Examine the effects of CET on fronto-temporal brain function. Functional MRI data using established executive and social cognition paradigms will be collected at baseline, 9, and 18 months along with cognitive and functional outcome data. It is hypothesized that CET patients will demonstrate enhanced fronto-temporal brain activity during these tasks relative to EST (see Section 3C.6.2 for specific predictions), and that this enhanced brain activity will be a mechanism of cognitive and functional improvement. Changes in fronto-temporal functional connectivity and their relations with improved brain structure and cognition will also be explored; and Aim #3: Examine the durability of CET effects on fronto-temporal brain structure and function, cognition, and functional outcome at 1 year post-treatment. Identical neuroimaging, cognitive, and behavioral data will be collected as those assessed during active treatment. It is hypothesized that the differential neurobiologic benefits of CET relative to EST observed in Aims 1 and 2, and the cognitive and functional benefits of CET observed during active treatment will be sustained 1 year post-treatment.

Exploratory Aim: Explore the effects of a fronto-temporal structural and functional reserve on CET treatment response. Moderator analyses will examine whether pre-treatment fronto-temporal structural and functional brain reserves (operationalized in Section 3C.8.2) predict larger cognitive and functional gains in CET. Exploratory analyses will also examine the degree to which later (18 mo) treatment improvement is dependent upon early (9 mo) neuroprotection and increased brain function, which may reflect plasticity.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they have:

1. a diagnosis of schizophrenia or schizoaffective disorder verified by the SCID (in our data patients with both conditions respond similarly to CET);
2. duration since first psychotic symptom of < 10 years;
3. stable positive symptoms based on medical record review and SCID for at least 2 months;
4. are currently maintained on and compliant with prescribed antipsychotic medication;
5. age 18-55 years;
6. significant social and cognitive disability based on the Cognitive Style and Social Cognition Eligibility Interview utilized in previous CET studies;
7. current IQ >= 80; and
8. the ability to read (sixth grade level or higher) and speak fluent English. This is a study of early course schizophrenia, not first-episode schizophrenia. A duration of illness since first psychotic symptom of < 10 years is adequate to define the early phase of the illness, particularly given that the average duration of untreated psychosis is a year or more. Eligibility criteria regarding IQ are justified from previous experience with CET indicating that individuals with severe mental incapacity are better served with less cognitively advanced programs.

Exclusion Criteria:

In order to avoid confounders likely to affect cognition and limit response to cognitive rehabilitation, we will exclude those with:

1. significant neurological or medical disorders that may produce cognitive impairment (e.g., seizure disorder, traumatic brain injury);
2. persistent suicidal or homicidal behavior;
3. a recent (within the past 3 months) history of substance abuse or dependence; and
4. any MRI contraindications such as ferromagnetic objects in the body.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Confirm the neuroprotective effects of CET on frontal and temporal brain structure | 18 months
  Aim #1: Confirm the neuroprotective effects of CET on frontal and temporal brain structure. Structural magnetic resonance imaging (MRI) assessments will be collected along with cognitive and functional outcome data at baseline, 9, and 18 months. It is hypothesized that patients treated with CET will demonstrate decreased loss of frontal and temporal gray matter relative to EST, and that this neuroprotection will be a mechanism of cognitive and functional improvement.
Examine the effects of CET on fronto-temporal brain function. | 18 Months
  Aim #2: Examine the effects of CET on fronto-temporal brain function. Functional MRI data using established executive and social cognition paradigms will be collected at baseline, 9, and 18 months along with cognitive and functional outcome data. It is hypothesized that CET patients will demonstrate enhanced fronto-temporal brain activity during these tasks relative to EST (see Section 3C.6.2 for specific predictions), and that this enhanced brain activity will be a mechanism of cognitive and functional improvement.
Examine the durability of CET effects on fronto-temporal brain structure and function, cognition, and functional outcome at 1 year post-treatment | 1 year post-treatment
  Aim #3: Examine the durability of CET effects on fronto-temporal brain structure and function, cognition, and functional outcome at 1 year post-treatment. Identical neuroimaging, cognitive, and behavioral data will be collected as those assessed during active treatment. It is hypothesized that the differential neurobiologic benefits of CET relative to EST observed in Aims 1 and 2, and the cognitive and functional benefits of CET observed during active treatment will be sustained 1 year post-treatment.

SECONDARY OUTCOMES:
Explore the effects of a fronto-temporal structural and functional reserve on CET treatment response. | 18 Months
  Exploratory Aim: Explore the effects of a fronto-temporal structural and functional reserve on CET treatment response. Moderator analyses will examine whether pre-treatment fronto-temporal structural and functional brain reserves (operationalized in Section 3C.8.2) predict larger cognitive and functional gains in CET. Exploratory analyses will also examine the degree to which later (18 mo) treatment improvement is dependent upon early (9 mo) neuroprotection and increased brain function, which may reflect plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Matcheri Keshavan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Psychiatry Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Keshavan MS, Hogarty GE. Brain maturational processes and delayed onset in schizophrenia. Dev Psychopathol. 1999 Summer;11(3):525-43. doi: 10.1017/s0954579499002199. PMID 10532623
- [Background] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824
- [Background] Insel TR. Translating scientific opportunity into public health impact: a strategic plan for research on mental illness. Arch Gen Psychiatry. 2009 Feb;66(2):128-33. doi: 10.1001/archgenpsychiatry.2008.540. PMID 19188534
- [Derived] Wojtalik JA, Mesholam-Gately RI, Hogarty SS, Greenwald DP, Litschge MY, Sandoval LR, Shashidhar G, Guimond S, Keshavan MS, Eack SM. Confirmatory Efficacy of Cognitive Enhancement Therapy for Early Schizophrenia: Results From a Multisite Randomized Trial. Psychiatr Serv. 2022 May;73(5):501-509. doi: 10.1176/appi.ps.202000552. Epub 2021 Sep 2. PMID 34470506
- [Derived] Hegde RR, Guimond S, Bannai D, Zeng V, Padani S, Eack SM, Keshavan MS. Theory of Mind impairments in early course schizophrenia: An fMRI study. J Psychiatr Res. 2021 Apr;136:236-243. doi: 10.1016/j.jpsychires.2021.02.010. Epub 2021 Feb 13. PMID 33621908
- [Derived] Guimond S, Ling G, Drodge J, Matheson H, Wojtalik JA, Lopez B, Collin G, Brady R, Mesholam-Gately RI, Thermenos H, Eack SM, Keshavan MS. Functional connectivity associated with improvement in emotion management after cognitive enhancement therapy in early-course schizophrenia. Psychol Med. 2022 Sep;52(12):2245-2254. doi: 10.1017/S0033291720004110. Epub 2020 Nov 13. PMID 33183362
- [Derived] Hegde RR, Kelly S, Lutz O, Guimond S, Karayumak SC, Mike L, Mesholam-Gately RI, Pasternak O, Kubicki M, Eack SM, Keshavan MS. Association of white matter microstructure and extracellular free-water with cognitive performance in the early course of schizophrenia. Psychiatry Res Neuroimaging. 2020 Nov 30;305:111159. doi: 10.1016/j.pscychresns.2020.111159. Epub 2020 Aug 14. PMID 32919288
- [Derived] Guimond S, Padani S, Lutz O, Eack S, Thermenos H, Keshavan M. Impaired regulation of emotional distractors during working memory load in schizophrenia. J Psychiatr Res. 2018 Jun;101:14-20. doi: 10.1016/j.jpsychires.2018.02.028. Epub 2018 Mar 2. PMID 29524918